CLINICAL TRIAL: NCT03930940
Title: Safey and Efficacy of Remote Ischemic Conditioning in Patient With Spontaneous Intracerebral Hemorrhage
Brief Title: Remote Ischemic Conditioning for Intracerebral Hemorrhage
Acronym: RICH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Heze Municipal Hospital (Other); The Sixth People's Hosptial of Hengshui (Unknown); Weihai Municipal Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RICH
Record Dates: First submitted 2019-04-20; First posted 2019-04-29 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Intracerebral Hemorrhage
Keywords: Spontenous intracerebral hemorrhage; Hemorrhage resolution; Remote ischemic conditioning; Neuroprotection
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): RIC treatment and regular treatment.
  Interventions: Device: remote ischemic conditioning; Other: Regular treatment
- Control group (Other): Regular treatment alone.
  Interventions: Other: Regular treatment

INTERVENTIONS:
Device: remote ischemic conditioning — RIC is a non-invasive therapy that performed by an electric autocontrol device with cuffs placed on arm and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 4 to 5 times.
  Arms: RIC group
Other: Regular treatment — Regular treatment is based on associated guidelines for ICH.

SUMMARY:
Spontaneous intracerebral hemorrhage (ICH) results from the rupture of small vessels damaged by chronic hypertension, amyloid angiopathy or other disease. Hematoma volume has been demonstrated to be strongly correlated with the severity of white matter injury and conditions in ICH patients. In the past decades, surgical clot evacuation and stereotactic or endoscopic clot aspiration with thrombolytic drugs have been investigated for the treatment of ICH, however, none of them have been demonstrated to be effective. As such, medical management remains the standard of care for most patients with ICH, leading to ICH as the least treatable form of stroke.

Remote ischemic conditioning (RIC) has been found to have neuroprotective effects by in patients with ischemic stroke. In addition, animal studies show that RIC is safe in ICH model and it could accelerate the absorption of hematoma. Therefore, the investigators plan to undertake this study to evaluate the safety of RIC in patients with ICH, and planned for future study to determine if treatment with RIC can improve the outcome of patients with ICH.

In this study, our main objectives are: 1) to evaluated the safety of RIC, by determining the treatment related adverse events, in patients with ICH; and 2) to determine the preliminary effects of RIC on hematoma absorption and cerebral edema.

The investigators hypothesize that RIC is well-tolerated and has minimal serious adverse effects in patients with ICH; and that treatment with RIC will accelerate the absorption of hematoma and improve patients' functional outcomes. Results of this study can potentially bring into account new means to improve the outcomes of ICH patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 and ≤80.
2. The diagnosis of ICH is confirmed by brain CT scan.
3. Hematoma volume of 10 to 30 ml.
4. Glasgow Coma Score (GCS)>8.
5. Starting RIC treatment between 24 and 48 hours of ictus.
6. Signed and dated informed consented is obtained.

Exclusion Criteria:

1. Patients with suspected secondary ICH related to tumor, coagulopathy, ruptured aneurysm or arteriovenous malformation, or venous sinus thrombosis.
2. ICH concomitant with subarachnoid hemorrhage or intraventricular hemorrhage. Planned surgical evacuation of hematoma prior to RIC.
3. Evidence of significant shift of midline brain structure (> 10 mm) or herniation on brain imaging.
4. Known pregnancy (or positive pregnancy test), or breast-feeding.
5. Concurrent participation in another research protocol for investigation of another experimental therapy.
6. Patients with a pre-existing neurological deficits (modified Ranks scale score >1) or psychiatric disease that would confound the neurological or functional evaluations.
7. Life expectancy of less than 90 days due to co-morbid conditions.
8. Severe hepatic and renal dysfunction.
9. Severe, sustained hypertension (SBP > 180 mmHg or DBP > 110 mmHg).
10. Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs.
11. Any condition which, in the judgment of the investigator, might increase the risk to the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, PhD, Principal Investigator — Xuanwu Hospital, Capital Medical Univeristy
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaibhav K, Braun M, Khan MB, Fatima S, Saad N, Shankar A, Khan ZT, Harris RBS, Yang Q, Huo Y, Arbab AS, Giri S, Alleyne CH Jr, Vender JR, Hess DC, Baban B, Hoda MN, Dhandapani KM. Remote ischemic post-conditioning promotes hematoma resolution via AMPK-dependent immune regulation. J Exp Med. 2018 Oct 1;215(10):2636-2654. doi: 10.1084/jem.20171905. Epub 2018 Sep 6. PMID 30190288
- [Background] Zhao W, Meng R, Ma C, Hou B, Jiao L, Zhu F, Wu W, Shi J, Duan Y, Zhang R, Zhang J, Sun Y, Zhang H, Ling F, Wang Y, Feng W, Ding Y, Ovbiagele B, Ji X. Safety and Efficacy of Remote Ischemic Preconditioning in Patients With Severe Carotid Artery Stenosis Before Carotid Artery Stenting: A Proof-of-Concept, Randomized Controlled Trial. Circulation. 2017 Apr 4;135(14):1325-1335. doi: 10.1161/CIRCULATIONAHA.116.024807. Epub 2017 Feb 7. PMID 28174194
- [Background] Zhao W, Zhang J, Sadowsky MG, Meng R, Ding Y, Ji X. Remote ischaemic conditioning for preventing and treating ischaemic stroke. Cochrane Database Syst Rev. 2018 Jul 5;7(7):CD012503. doi: 10.1002/14651858.CD012503.pub2. PMID 29974450
- [Background] Zhao W, Che R, Li S, Ren C, Li C, Wu C, Lu H, Chen J, Duan J, Meng R, Ji X. Remote ischemic conditioning for acute stroke patients treated with thrombectomy. Ann Clin Transl Neurol. 2018 Jun 6;5(7):850-856. doi: 10.1002/acn3.588. eCollection 2018 Jul. PMID 30009202
- [Background] Zhao W, Li S, Ren C, Meng R, Jin K, Ji X. Remote ischemic conditioning for stroke: clinical data, challenges, and future directions. Ann Clin Transl Neurol. 2018 Nov 15;6(1):186-196. doi: 10.1002/acn3.691. eCollection 2019 Jan. PMID 30656197
- [Derived] Ma H, Gu Y, Bian T, Song H, Liu Z, Ji X, Duan J. Dabigatran etexilate versus warfarin in cerebral venous thrombosis in Chinese patients (CHOICE-CVT): An open-label, randomized controlled trial. Int J Stroke. 2024 Jul;19(6):635-644. doi: 10.1177/17474930241234749. Epub 2024 Feb 26. PMID 38353219
- [Derived] Zhao W, Jiang F, Li S, Liu G, Wu C, Wang Y, Ren C, Zhang J, Gu F, Zhang Q, Gao X, Gao Z, Song H, Ma Q, Ding Y, Ji X; RICH-1 Investigators. Safety and efficacy of remote ischemic conditioning for the treatment of intracerebral hemorrhage: A proof-of-concept randomized controlled trial. Int J Stroke. 2022 Apr;17(4):425-433. doi: 10.1177/17474930211006580. Epub 2021 Apr 7. PMID 33739197
- [Derived] Zhao W, Jiang F, Li S, Wu C, Gu F, Zhang Q, Gao X, Gao Z, Song H, Wang Y, Ji X; RICH-1 Investigators. Remote Ischemic Conditioning for Intracerebral Hemorrhage (RICH-1): Rationale and Study Protocol for a Pilot Open-Label Randomized Controlled Trial. Front Neurol. 2020 Apr 28;11:313. doi: 10.3389/fneur.2020.00313. eCollection 2020. PMID 32411082